CLINICAL TRIAL: NCT01257074
Title: A Randomized, Double-Blind, to Compare Non-inferiority Efficacy and Safety of Penciclovir 10mg/g to Acyclovir 50mg/g in the Treatment of Recurrent Herpes Labialis.
Brief Title: Non-inferiority Comparison of Efficacy and Safety of Penciclovir 10mg/g to Acyclovir 50mg/g in the Treatment of Recurrent Herpes Labialis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PENEMS1010
Record Dates: First submitted 2010-12-06; First posted 2010-12-09 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Herpes Labialis
Keywords: Herpes Simplex
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex | interventions — Acyclovir; penciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug 1 (Experimental): Penciclovir 10mg/g
  Interventions: Drug: Penciclovir 10mg/g
- Drug 2 (Active Comparator): Acyclovir 50mg/g
  Interventions: Drug: Acyclovir 50mg/g

INTERVENTIONS:
Drug: Acyclovir 50mg/g — Cream, dose 5 times daily during 5 days
  Arms: Drug 2
Drug: Penciclovir 10mg/g — Cream, dose 5 times daily during 5 days
  Arms: Drug 1

SUMMARY:
Herpes labialis is the most common recurrent manifestation of herpes simplex. The purpose of this study is to check the non-inferiority efficacy and safety of penciclovir 10mg/g as treatment for Herpes Labialis in comparison to acyclovir 50mg/g.

DETAILED DESCRIPTION:
Study design:

• Double blinded non-inferiority prospective parallel-group, intend to treat trial.

Study design:

* Experiment duration: 10 days
* 3 visits (days 1,5 and 10)
* Erythema, papule, vesicle, ulcer, crust and healed skin evaluation
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the study procedures agree to participate and give written consent.
2. Patients with clinical diagnosis of recurrent herpes labialis and are in the prodromal period (stinging, itching, burning and erythema) at the onset of signs / symptoms in the last 12-24 hours;
3. No history of reaction to topical products;

Exclusion Criteria:

1. Pregnancy or risk of pregnancy.
2. Lactation
3. Use of anti-inflammatory or immunosuppressive drugs (last 30 days prior to the study.)
4. Sunlight over exposure in the last 15 days.
5. Any pathology or past medical condition that can interfere with this protocol.
6. AINH use, hormonal anti-inflammatory, analgesic and immunosuppressive drugs (in the last 30 days and during the study);
7. Patients with immunodeficiency and/or immunosuppressive disease;
8. Sunlight exposure in the last 15 days;
9. Hypersensitivity to components of the formula;
10. Other conditions deemed reasonable by the medical investigator as to the disqualification of the individual from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy will be evaluated by the proportion of subjects with non herpes labialis manifestation | Day 10
  Symptoms evaluated: erythema, papule, vesicle, ulcer, crust, or healed skin.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Addor, MD, Principal Investigator — Medcin Instituto da Pele Ltda
Locations (1):
- Flavia Addor, São Paulo, São Paulo, Brazil